## **Cover Sheet**

Study Title: MUCINEX for Treatment of Filamentary Keratitis

NCT No: NCT02859246

Date: 7/21/2019

## Statistical Analysis Performed



## Statistical Test of Hypothesis

added oral quaifenesin as a new treatment at baseline and patients who re-

ceived oral guaifenesin and an increase in topical corticosteroids simulta-

We calculated the difference in the mean number of filaments and OSDI score between baseline and follow-up visits and evaluated their change over time. We used the pairedsample Wilcoxon signed-rank test if data did not follow a normal distribution and the paired Student t-test in the case of normally distributed data. For all the analyses we considered the average value of both eyes for all variables with the exception of symptom scores (OSDI), which were considered per patient. Data are presented as the mean ± standard deviation (SD), a range for continuous variables, and percentages for categorical variables. A twotail P value of less than 0.05 was considered statistically significant in all statistical tests. The statistical analysis was performed using STATA 13.0 (StataCorp, College Station, TX).

guaifenesin and an increase in topical corticosteroids simultaneously